CLINICAL TRIAL: NCT00380913
Title: A Multicenter Trial Evaluating the Efficacy of Cesamet™ for the Symptomatic Treatment of Pain in Patients With Diabetic Peripheral Neuropathy
Brief Title: Evaluation of the Efficacy of Cesamet™ for the Treatment of Pain in Patients With Diabetic Peripheral Neuropathy
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: NEMA Research, Inc. (Industry)
Responsible Party: Joseph Pergolizzi, MD, NEMA Research
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CB1 Study 001
Record Dates: First submitted 2006-09-25; First posted 2006-09-27 (Estimated); Last update posted 2008-02-15 (Estimated); Status verified 2008-02

CONDITIONS: Diabetic Neuropathies
MeSH Terms: conditions — Diabetic Neuropathies | interventions — nabilone

INTERVENTIONS:
Drug: Cesamet™ (nabilone)

SUMMARY:
This study was designed to evaluate the safety and efficacy of Cesamet™ in controlling pain in subjects experiencing pain due to diabetic peripheral neuropathy.

DETAILED DESCRIPTION:
The purpose of this study is to determine the safety and efficacy of Cesamet™ in the symptomatic treatment of pain due to diabetic peripheral neuropathy.

This is a phase IV, multi-center, open label outpatient clinical trial evaluating Cesamet™ treatment for control of pain due diabetic peripheral neuropathy. The study has two phases: a Pretreatment Phase and a Treatment Phase.

ELIGIBILITY:
Inclusion Criteria:

* Patients with diabetic peripheral neuropathic pain
* Chronic daily pain present for at least 2 months
* On stable analgesic regimen for one month
* Baseline pain score greater than 40mm on a visual analog scale

Exclusion Criteria:

* Hypersensitivity to compounds in study drug or similar drugs
* Pregnant or lactating females
* Drug or alcohol abuse
* Unstable medical condition

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 23 (Estimated)
Dates: Start 2006-09; Primary Completion 2007-10 (Actual); Study Completion 2007-10 (Actual)

PRIMARY OUTCOMES:
The Average Pain Score at target site.

SECONDARY OUTCOMES:
The Worst Pain Score at target site.
The Pain at Night Score at target site.
Quality of Life measures
Patient satisfaction with treatment
Safety will be assessed through the collection of AEs and vital signs.

CONTACTS AND LOCATIONS:
Overall Officials: Joseph V Pergolizzi, MD, Principal Investigator — NEMA Research, Inc.; Charlotte Richmond, PhD, Study Director — Nema Research
Locations (4):
- United States (4):
  - South Florida Medical Research, Aventura, Florida
  - Sunrise Clinical Research, Inc., Hollywood, Florida
  - Naples Anesthesia and Pain Associates, Naples, Florida
  - Lazlo Mate, MD, West Palm Beach, Florida

REFERENCES:
- See also: Nema Research website — http://www.nema.net